CLINICAL TRIAL: NCT01856205
Title: A Randomized Double Blind Placebo Controlled Trial to Assess the Safety and Efficacy of Intravenous Immunoglobulin (IVIG) in Children With Japanese Encephalitis in Nepal
Brief Title: Safety and Efficacy Study of Intravenous Immunoglobulin to Treat Japanese Encephalitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Kanti Children's Hospital (Other); B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Ajit Rayamajhi, Clinical Research Fellow (PhD Student), University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVIG607
Record Dates: First submitted 2013-05-05; First posted 2013-05-17 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Japanese Encephalitis
Keywords: Japanese Encephalitis, Randomized Controlled Trial, intravenous immunoglobulin, safety, efficacy, Nepal
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IVIG in JE (JE-positive) (Placebo Comparator): We randomly allocated patients to treatment with IVIG or placebo. Children received either saline or intravenous immunoglobulin (IVIG) [ImmunoRel™ (batch 20081217)] at a dose of 400mg/kg/day for 5 days or an equivalent volume of 0.9% normal saline given intravenous at the rate of 0.01 to 0.02 ml/kg body weight/minute. All investigators, care providers and participants were blinded of the study drug. A second sealed envelope was kept with the patient's notes in case a physician urgently needed to know which drug a patient had received.
  Interventions: Drug: Intravenous immunoglobulin [ImmunoRel™ (batch 20081217)]
- IVIG in Non-JE(JE-negative) (Placebo Comparator): We randomly allocated patients to treatment with IVIG or placebo. Children received either saline or intravenous immunoglobulin (IVIG) [ImmunoRel™ (batch 20081217)] at a dose of 400mg/kg/day for 5 days or an equivalent volume of 0.9% normal saline given intravenous at the rate of 0.01 to 0.02 ml/kg body weight/minute. All investigators, care providers and participants were blinded of the study drug. A second sealed envelope was kept with the patient's notes in case a physician urgently needed to know which drug a patient had received.
  Interventions: Drug: Intravenous immunoglobulin [ImmunoRel™ (batch 20081217)]

INTERVENTIONS:
Drug: Intravenous immunoglobulin [ImmunoRel™ (batch 20081217)] — IVIG group received 400mg/kg/day intravenous at the rate of 0.01 to 0.02 ml/kg body weight/minute for 5 days or appearance of side effect or adverse events.
  Placebo group received 0.9% saline intravenous at similar rate.

SUMMARY:
Japanese encephalitis is caused by a viral infection of the brain transmitted by the bite of an infected mosquito. Patients with Japanese encephalitis can rapidly develop worsening conscious level and seizures. Around a third will die from the infection and half of survivors have serious long-term neurological disability. The majority of those affected are children. There are many causes of viral encephalitis, however Japanese encephalitis virus is the most common cause worldwide with over 60,000 cases annually. It occurs over much of Asia and the geographical range is expanding. There is no specific treatment for Japanese encephalitis virus, although several have been trialed. In this study we examined the effect of a new treatment, called intravenous immunoglobulin, on children with Japanese encephalitis in Nepal. Prior studies have suggested intravenous immunoglobulin may neutralize Japanese encephalitis virus and suppress damaging inflammation in the brain. It has previously been used in individual cases but never examined in a randomized trial. There was recently a trial of IVIG in West Nile encephalitis in the United States, in which Professor Solomon was on the Scientific Advisory Committee. In this study we will look if intravenous immunoglobulin is safe in this context, and that this treatment may alter the way the immune system manages the infection. Therefore, in this pilot study we will test the hypothesis that IVIG can be safely given to children with suspected JE, with no increased risk of serious adverse events compared with placebo. The aim of this proposal is to conduct a pilot safety and tolerability randomized placebo controlled trial of intravenous immunoglobulin (IVIG) in patients with Japanese encephalitis, to explore the relationship between JEV viral load, pro-inflammatory markers called cytokines and blood brain barrier markers, and the effect of IVIG on these relationships.

DETAILED DESCRIPTION:
Japanese encephalitis (JE) is the most important epidemic encephalitis worldwide, causing approximately 35-50,000 cases and 10-15,000 deaths annually. Half of the survivors have severe neuropsychiatric sequelae, posing a large socio-economic burden on communities that can ill afford it. JE virus (JEV, genus flavivirus, family Flaviviridae) has a 50 nm lipoprotein envelope surrounding a nucleocapsid comprised of core protein and 11 KB of single-stranded positive-sense RNA. The genome has 5' and 3' untranslated regions (UTR), and a single open reading frame encoding genes for three structural proteins (core - C, pre-membrane - prM and envelope - E) and 7 non-structural (NS) proteins. The E protein is critical for viral attachment and entry into cells, and along with NS1 and NS3 is a major target of the immune response.

JEV is an arthropod-borne virus (arbovirus), transmitted in an enzootic cycle between birds, pigs and other vertebrates by mosquitoes, especially Culex species. Almost all of the population in affected parts of Asia is infected by early adulthood, but only a small proportion (about 1 in 300) develops clinical features. These may range from a non-specific febrile illness to a severe meningoencephalitis, in which seizures and clinical signs of raised intracranial pressure are common, and carry a poor prognosis. In addition JEV causes a poliomyelitis-like flaccid paralysis. The distribution of the four genotypes of JEV across Asia was thought to explain the clinical epidemiology, but is now thought to be a reflection of the virus' origin in Southeast Asia, and spread from here. However subtle differences in the genome may be important in determining neurological presentations of flaviviruses.

Although there are vaccines against JEV, they are not available for many of the people that need them, because of issues over cost and production. Progress is being made to overcome these difficulties, and newer vaccines are being used increasingly. In fact Nepal has been at the forefront of the use of a single dose of live attenuated SA14-14-2 vaccine for JE. However, continues to spread across Asia, and there is no treatment. Interferon-α (IFN-α), which is produced as part of the innate response to JEV infection, and which has antiviral activity against the virus, was thought to be the most promising treatment. However, a randomized placebo-controlled trial showed recombinant IFN-α2a at 10 million units/m2/day did not improve the outcome. The pathogenesis of JE is incompletely understood, but by comparison with other positive sense RNA viral encephalitides, is likely to involve a mixture of viral cytopathology and immunopathology .The role of steroids in JEV has been examined in one randomized-placebo controlled trial in Thailand, which failed to show any benefit.

IVIG currently offers one of the best possibilities for improving the outcome in JE. It has been used presumptively in patients with flavivirus encephalitis, including JE, and is postulated to act in two ways: IVIG produced in countries where flaviviruses are endemic contains high titers of specific neutralizing antibody, because most of the population have been exposed to the virus, and thus have antibodies. In addition IVIG has non-specific anti-inflammatory properties, particularly through the suppression of pro-inflammatory cytokines (e.g. in Kawasaki disease). We aim to examine the role of IVIG in JE, and also look at its effects on pro-inflammatory cytokines.

The role of antibody in protection against severe disease in Japanese encephalitis: The humoral immune response in JE has been well characterized. When disease is due to primary infection (i.e. when JEV is the first flavivirus with which an individual has been infected) a rapid and potent IgM response occurs in serum and CSF within days of infection. By day 7 most patients have elevated titers. Attempts to isolate virus are usually negative in such patients. However, the failure to mount an IgM response is associated with positive virus isolation and a fatal outcome. Antibody to JEV probably protects the host by restricting viral replication during the viraemic phase, before the virus crosses the blood brain barrier. Evidence from other flaviviruses suggests it may also limit damage during established encephalitis by neutralizing extracellular virus and facilitating lysis of infected cells by antibody-dependent cellular cytotoxicity.

In surviving patients immunoglobulin class switching occurs, and within 30 days most have IgG in the serum and CSF. Asymptomatic infection with JEV is also associated with elevated IgM in the serum, but not CSF. In patients with secondary infection (i.e. those who have previously been infected with a different flavivirus, for example dengue infection, or yellow fever vaccination) there is an anamnastic response to flavivirus group common antigens. This secondary pattern of antibody activation is characterized by an early rise in IgG with a subsequent slow rise in IgM.

Inflammation in Japanese encephalitis: At autopsy in JE, the brain is usually edematous, with congestion of the parenchyma . Cerebellar and uncal herniation are common. Histopathologically JE is characterized by perivascular inflammation with recruitment of macrophages, neutrophils and lymphocytes. The basal ganglia and anterior horns cells of the spinal cord are particularly affected, providing a pathological correlate for the Parkinsonism, and poliomyelitis-like flaccid paralysis, which may be seen. Viral antigen is predominantly in neurons although microglial cells, astrocytes and vascular endothelial cells are also infected. When survival is prolonged beyond 7 days acellular necrotic zones are seen, usually in the region of small or medium sized arteries which are surrounded by edema.

Immunopathology in Japanese encephalitis: The pathogenesis of JE is incompletely understood, but available evidence indicates that, as with a number of other positive sense RNA viral encephalitides including lymohoctyic chorio meningitis virus (LCMV) in mice Sindbis virus, dengue virus, yellow fever virus and West Nile virus, there is immune-mediated damage as well as viral cytopathology.

Pro-inflammatory cytokine responses in Japanese encephalitis: As detailed below under Preliminary Studies, there is accumulating evidence that the pro-inflammatory cytokine response may make an important contribution to immunopathology in JE. Among cytokines studied, interleukin (IL)-6, IL-8 chemokine (CXC motif) ligand (CXCL-8), and tumor necrosis factor (TNF)- α appear to be associated with a fatal outcome. There is also new evidence on the importance of other cytokines and chemokines in encephalitis caused by other flaviviruses, particularly West Nile virus. There are several mechanisms by which the pro-inflammatory response may be deleterious. Recent studies have shown IL-6, which is produced by neurons, microglia, astrocytes and recruited macrophages in response to viral CNS infection, causes an increased permeability of the blood brain barrier (BBB), which leads to interstitial cerebral edema, and raised intracranial pressure. TNF-α is produced by microglia, astrocytes and macrophages. Its multiple pro-inflammatory properties include upregulation of class I and II MHC expression, upregulation of cellular adhesion molecules, increased permeability of the BBB, and upregulation of inducible nitric oxide synthase (iNOS), leading to the production of nitric oxide (NO). At high concentrations NO is directly toxic to CNS cells, causing oxidative damage, and apoptosis. Recent evidence suggests that the early cytokine and chemokines responses may also be important in determining whether the virus even gains entry across the blood brain barrier to enter the CNS. In one study of West Nile virus infection, mice deficient in Toll-like receptor 3(Tlr3), which recognizes viral double stranded RNA, were relatively resistant to lethal infection. This was associated with reduced cytokine production (particularly TNF-α and IL-6), and increased viral load in the periphery, compared to wild type mice. TNF-α receptor 1 signaling was found to be vital for blood brain barrier compromise upon Tlr3 stimulation by the virus. In addition to affecting virally-infected cells, the inflammatory response in the CNS may also damage non-infected cells to cause bystander cell death. The importance of the chemokine receptor CCR5, and its ligand CCL5 (also known as RANTES, regulated on activation, normally T cell expressed and secreted) in CNS inflammation caused by flaviviruses was shown recently by their prominent up-regulation in a mouse model of West Nile virus infection. This was associated with CNS infiltration of CD4+ and CD8+ T cells, Natural killer (NK)1.1+ cells and macrophages expressing the receptor. The significance of CCR5 in pathogenesis was established by mortality studies in which infection of CCR5-/- mice was rapidly and uniformly fatal. Importantly, our recent study (see below) found that CCL5 was also elevated in the plasma of humans with JE, where higher levels were associated with a fatal outcome.

Although clinical studies in humans with JE, and parallel studies in animal models of flavivirus encephalitis suggest elevated pro-inflammatory cytokines appear to be important and associated with a bad outcome in JE, it is not clear whether control of this strong pro-inflammatory response will improve the outcome. We will conduct a pilot double-blind placebo-controlled study on safety, tolerability and immunological markers of efficacy of IVIG in children with JE in Nepal, followed by a larger efficacy study.

Preliminary studies: Professor Solomon has been studying JE and related flaviviruses since 1994. With the support of his group and collaborators, he has shown that JEV is the most important cause of viral encephalitis in Vietnam, as it is in most of South and Southeast Asia. He showed that seizures and raised intracranial pressure are common clinical manifestations of infection. In collaboration with colleagues in Malaysia he developed and field-tested a simple rapid diagnostic test for diagnosing JE in the rural settings where it occurs. This test was also able to distinguish JE from dengue - a related flavivirus that circulates in Asia. Although dengue is better known as a cause of hemorrhagic disease, Prof Solomon and his team showed that it is also an important cause of neurological disease. Prof Solomon also showed that as well as presenting with encephalitis, JEV can present with a poliomyelitis-like acute flaccid paralysis, which has also more recently been recognized in adults infected with West Nile virus. Based on in vitro and in vivo data, together with phase I/II studies in humans, Prof Solomon conducted a randomized placebo controlled trial of interferon α-2b in children with JE (the only antiviral trial ever conducted for JE). However the study showed that it did not improve the outcome. To begin exploring the possible contribution of viral genetic diversity to the clinical epidemiology of JE, Prof Solomon examined the molecular evolution of the virus across Asia, and showed that the virus probably originated in the Indonesia and Malaysia region, and evolved here into the different genotypes, the most recent of which subsequently spread across Asia.

The Liverpool group has more recently begun examining inflammation in JE. A recent pathological study in humans and a mouse model confirms the importance of the inflammatory response, and suggests there may be damage to the vascular endothelium. A study of pro-inflammatory and anti-inflammatory cytokines in humans with JE has shown that CSF levels of interleukin(IL)-6, tumor necrosis factor (TNF)-α, interferon (IFN)-α and the chemokine CXCL8 (IL-8) were higher in patients who died than in those who survived. IFN-γ and nitric oxide (NO) were also detected in the CSF of fatal cases and survivors. These findings extend the observations of other investigators on TNF-α and CXCL8 indicating a strong pro-inflammatory response in JE is associated with a poor outcome. It was also shown that CCL5 (RANTES) is expressed in the plasma of humans with JE, and that high plasma levels are associated with fatal disease. Clinical data from other flavivirus encephalitides support the concept that inflammation may contribute to the pathogenesis. For example, immunosuppressed transplant patients infected with West Nile virus develop CNS disease later than immunocompetent patients. Cytokines do not act in isolation, and indeed the pluripotency and redundancy of biological response is one of their characteristic features. Recent microarray experiments show a wide range of molecules are upregulated in CNS inflammatory conditions. In addition the Liverpool group has studied the relationship between antibody responses and outcome. Along with other investigators, we have shown that the presence of antibody in the serum and CSF is associated with survival.

JE in Nepal: Japanese encephalitis was first recorded in Nepal in 1978 and is currently endemic in 24 districts. Since its first appearance there have been over 26,667 cases and 5381 deaths. The early mortality figures were quoted at up to 60%, but more recently they have improved to approximately 20% in those under 15 years. The morbidity is thought to be around 50%. As a result of concern about the disease, there was immunization against JE in 1999 in 3 districts, this has now been extended to cover the majority of the affected districts. In addition the Government vaccinated around 200 000 pigs in the Terai zone in 2001. Despite these successes there are still ongoing cases of JE. In 2006 there were 292 confirmed cases and 1481 AES cases of unknown etiology. These figures may under represent the actual numbers of cases due to logistical issues, deaths before hospital admission, and difficulties in confirming the diagnosis of JE with paired sera and CSF samples. Recent serosurveillance in the animal hosts for JE in Nepal clearly shows the virus is still present in the wild and is likely to remain. Seroprevalence was 48% (102/212), in pigs, 27% (15/56) in ducks and 50% (6/12) in horses from a total of 280 sera collected from 10 districts of which 44% were positive overall. Hence, JE is still a major public health problem in Nepal, and there is a pressing need to develop better treatments. Currently IVIG is used in Nepal to treat a range of pediatric conditions, including Guillain-Barré syndrome, idiopathic thrombocytopenic purpura.

Rationale for use of IVIG in JE: There is currently no antiviral or immunomodulatory treatment for JE or indeed any flavivirus encephalitis. As outlined above, the only trials conducted, using interferon alpha, and using dexamethasone, failed to show any benefit. Based on data in preclinical studies, and observational studies in humans (see below), IVIG currently offers the best hope for treatment, through its antiviral and anti-inflammatory properties.

Established pediatric uses of IVIG: IVIG has been established as the standard treatment for a number of childhood immune mediated diseases including Guillain-Barré syndrome, Kawasaki's disease, immune thrombocytopenia and Dermatomyositis. In Kawasaki disease, T cell and B cell activation is down regulated by IVIG. In thrombocytopenic purpura blockade of FCγ receptors is thought to be important, which may result in down regulation of secretory cytokines. In Guillain-Barré syndrome and dermatomyositis inhibition of complement binding and prevention of membranolytic attack complex formation are possible mechanisms of IVIG action. In addition, IVIG has been employed in the treatment and prophylaxis of a number of childhood viral infections where the neutralizing antibodies in the IVIG were thought to be important. IVIG has been used to treat, and later to provide prophylaxis, for children with hypo- or agammaglobulinamia with chronic enteroviral meningoencephalitis. Importantly, children with X-linked agammaglobulinaemia and with enteroviral meningoencephalitis treated with intensive and prolonged IVIG therapy have achieved long-lasting clinical and viral remission (negative CSF viral culture and PCR). However, the patients relapsed when IVIG was tapered, indicating a major beneficial role of IVIG in this condition. IVIG infusion in infants and children with AIDS treated with zidovudine therapy has been shown to reduce the risk of serious bacterial infections (16.9% IVIG group vs 24.3% placebo group (relative risk, 0.60; 95 percent confidence interval, 0.35 to 1.04; p = 0.07). In respiratory syncytial virus (RSV) infections immunoglobulin therapy has been shown to be safe and generally well tolerated in a randomized controlled trial (RCT) involving 102 previously healthy children, though the beneficial effect of reducing hospitalization and intensive care unit day were marginal in children with severe disease. Other established indications for passive immunization with IVIG include parvovirus B19 infection.

Use of IVIG in flavivirus encephalitis: There is strong evidence to suggest that JEV, like other neurotropic flaviviruses, may be more susceptible to antibody-mediated, rather than cell-mediated immune responses. For JEV, and other neurotropic flaviviruses, clearance of virus is not dependent on cytolytic T cell activity, in contrast to non-neurotropic viruses. Neurons, as terminally differentiated cells, do not express MHC-1, which would subject them to lysis by CD8 T cells and non-replacement. Animal data support the importance of antibody mediated immunity. In one study, Konishi et. al. immunized mice with plasmid DNAs encoding JEV proteins that induce neutralizing antibody responses or cytotoxic T lymphocyte responses, and then challenged with lethal intraperitoneal doses of virus. They showed that neutralizing antibody prevents virus dissemination from the peripheral site to the brain, and that antibody-mediated mechanisms of protection were more efficient than the cytotoxic T cell responses. These findings supported earlier work showing that anti-envelope protein antibodies, are the most critical protective component in a JEV challenge model, and more recent passive antibody transfer experiments. In vitro work in mice shows a protective role for IVIG given prophylactically to prevent the flavivirus causing tick borne encephalitis and a protective effect when used as a treatment. In work by several different groups, use of IVIG containing specific anti West Nile Virus antibody during the viraemic phase, before the virus had entered the CNS, showed a dramatic 100% survival. Similar work with Tick borne encephalitis had a 100% effect on survival. There are now good data that in animal models of flavivirus encephalitis, peripheral administration of antibody neutralizes virus even after it has entered the central nervous system.

Clinical Data: Because of the of preclinical data supporting a role for antibody treatment in flavivirus encephalitis, antibody treatment (in the form of IVIG) has also been used on a compassionate basis in JE, and West Nile encephalitis. In addition IVIG is currently being investigated for West Nile encephalitis in a National Institutes of Health (NIH) sponsored randomized placebo controlled trial in the United States (for which Prof Solomon is on the Scientific Steering Committee).

IVIG was used in a 49 year old traveler returning from Vietnam who presented with JE to an Italian hospital. IVIG has also been used to treat West Nile virus infections in five patients in Israel and three in the United States. IVIG was also assessed in a placebo controlled trial for West Nile virus infection in the United States with no serious adverse effects of the drug.

Rationale for Dose: The most commonly used dose of IVIG is 2g/kg, either given as a single infusion, or divided as 400mg/kg for five days. In Kawasaki disease 2g/kg as a single ten hour infusion is well tolerated, and was shown to be the most effective regime. In Guillain-Barré syndrome in children and adults the drug is most often given over 5 days, and this is the regime that has been used in patients with flavivirus encephalitis, and will be used in this study.

Drug and Intervention: Children that meet the entry criteria will be randomly assigned to receive IVIG, (Reliance Biophamaceuticals Pvt. Ltd.) at a dose of 400mg/kg/day for 5 days, or an equivalent volume of 0.9% normal saline, using an established technique for giving fluid treatment in a double blind manner.

Drug Presentation: We will use Immunorel™ intravenous immunoglobulin, which is produced by Reliance Biophamaceuticals Pvt. Ltd., and manufactured in China and is available through the Yetichem Pharmacy, Sundhara, Kathmandu and Shriran Pharmacy, Maharajgunj, Kathmandu. This is the IVIG product currently used most often in Nepal.

As for most other parts of Asia, the seroprevalence of JE in China is high. By age 10, approximately one third of children have neutralizing antibodies to JEV, and by adulthood, the majority of the population has been exposed. There are extensive data showing that IVIG from areas where flaviviruses are endemic contains significant amounts of neutralizing antibody. For example for IVIG from Israel contains moderate to high levels of neutralizing antibody to West Nile Virus. Even though West Nile virus has only circulated in the United States for a few years, high levels of neutralizing antibody have been found in some IVIG lots.

Anti-JEV neutralizing antibody in IVIG from Asia: We have recently examined the neutralizing antibody titres in a range of IVIG products from India and China, using the plaque reduction neutralization assay (PRNT)50. In this study we found that IVIG from the UK, contained no antibody, and serum from a laboratory worker who had been vaccinated against JEV contained a small amount of neutralizing antibody. In contrast IVIG manufactured by Bharrat, Hualan, Sichun and Reliance companies all had neutralizing antibody titres of greater than 1 in 400, with Reliance having the greatest titre, at nearly 1 in 750.

Immunorel™ is packed in clear and colorless vials and comes in 2 pack sizes, each containing IVIG at a dose of 0.05g/ml (ie 50mg/ml). The available vials are, 50ml (containing 2.5g), and 100ml (5.0g).

Children will thus receive 400mg/kg/day of IVIG which is equivalent to 8mls/kg/day of Immunorel™ solution, or 8ml/kg/day of 0.9% normal saline.

Pharmacokinetics: Distribution studies have been done with a range of IVIG preparations. In a study of patients who developed aseptic meningitis (as a complication of the infusion), after receiving 2 g/kg intravenously in 2 divided doses, the serum level increases fivefold and then declines by 50% over the next 72 hours as extravascular redistribution took place. By 21- 28 days, pretreatment levels were reached. The half-life was 18-32 days, and was similar to native immunoglobulin. In the first 48 hours after the infusion the CSF concentration increased 1.5 to 7-fold but returned to normal within a week. CNS penetration may be expected in patients with viral meningoencephalitis or even encephalomyelitis as there will be a break down of the blood-brain-barrier. Metabolism of IVIG takes place in the cells of the reticuloendothelial system where immunoglobulins and immunoglobulin complexes are broken down.

Studies with Immunorel® in normal subjects showed that peak serum concentrations occur immediately after intravenous injection, and are dose related. Within 24 hours up to 30% of a dose may be removed by catabolism and distribution. Data concerning distribution suggest that IVIg distributes throughout intravascular (60%) and extravascular (40%) spaces. The serum half life of immunoglobulin ranges between 21 and 29 days.

Reaction Associated with Intravenous Immunoglobulin: Reactions to intravenous immunoglobulin tend to be related to the infusion rate and are most likely to occur during the first hour of the infusion. We will monitor the patient's vital signs and general status regularly throughout the infusion. The types of reactions that have been reported include abdominal pain, headache, chest-tightness, facial flushing or pallor, hot sensations, dyspnoea, non-urticarial skin rash, itching, hypotension, nausea or vomiting. Should any of these reactions develop during infusion of IVIG, the infusion will be temporarily stopped until the patient improves clinically (5 to 10 minutes) and then cautiously recommenced at a slower rate. Some patients may develop delayed adverse reactions to IVIG such as nausea, vomiting, chest pain, rigors, dizziness or aching legs. These adverse reactions occur after the infusion has stopped but usually within 24 hours. True hypersensitivity reactions to IVIG such as urticaria, angioedema, bronchospasm or hypotension occur very rarely. Should an anaphylactic reaction develop after IVIG, the infusion will be stopped and treatment instituted with adrenaline, oxygen, antihistamine and steroids. Hemolytic anemia and neutropenia have been reported in rare instances in association with IVIG treatment. Mild and moderate elevations of serum transaminases (AST, ALT, gamma GT) have been observed in a small number of patients given IVIG. Such changes were transient and not associated with the transmission of hepatitis. Rare complications an aseptic meningitis syndrome (AMS), thrombophlebitis, renal dysfunction and acute renal failure have occurred in patients receiving IVIG. Liver and renal function will be monitored during the study.

Reactions Associated with Immunorel™:

i. Primary Immune Deficiency: In patients with immunodeficiency syndrome receiving IVIG at a monthly dose of 400 mg/kg body weight, the reactions reported have been malaise, feeling of faintness, fever, chills, headache, nausea, vomiting, chest tightness, dyspnoea and chest, back or hip pain. Mild erythema at the infusion site has also been reported in some cases.

ii. Idiopathic Thrombocytopenic Purpura (ITP): In the treatment of adult and paediatric patients with ITP at a dose of 400 mg/kg body weight, the systemic reactions were observed only in less than 3% of the patients. The other symptoms which were all mild and transient include chest tightness, a sense of tachycardia and a burning sensation in the head. At a dose of 1000 mg/kg body weight either as a single dose or as two doses on consecutive days in the treatment of adult and paediatric patients with ITP. Adverse reactions have been noted only in less than 10% of the patients.

iii. Bone Marrow Transplantation: At a dose of 500 mg/kg body weight 7 days and two days before transplant and weekly through day 90 post-transplant, adverse reactions were reported in less than 7% of the patients. All reactions were classified as mild which include headache, flushing, fever and slight back discomfort.

iv. Renal: Increases in creatinine and blood urea nitrogen (BUN) may be seen as soon as one to two days after an infusion. Progression to oliguria or anuria may require dialysis. Severe occasional adverse events have been reported following IVIG therapy include: acute renal failure, acute tubular necrosis, proximal tubular nephropathy, and osmotic nephosis. Correction of volume depletion by using appropriate fluids prior to initiation of IVIG therapy is therefore essential. Measurement of blood urea nitrogen (BUN) and /or serum creatinine should be performed prior to initial infusion of IVIG and again at appropriate intervals afterwards, with monitoring of urine output.

iv. General: Reactions to IVIG are related to the rate of infusion. Very rarely an anaphylactoid reactions may occur in patients with no prior history of severe allergic reactions to either intramuscular or intravenous immunoglobulin.

Mutagenicity, Carcinogenicity and Impairment of Fertility: Animal reproduction studies have not been conducted with Gamma IV™. Hence it is not known whether IVIG can cause fetal harm when administered to pregnant woman or can affect the reproduction capacity.

Interactions with Other Drugs: The interaction of IVIG with other drugs has not been established in appropriate studies. Passively acquired antibody can interfere with the response to live, attenuated vaccines. Therefore, administration of such vaccines, e.g. poliomyelitis or measles, will be deferred until approximately six months after IVIG infusion. By the same token, immunoglobulins should not be administered for at least two weeks after a vaccine has been given.

Contraindications: IVIG is contraindicated in individuals who are known to have an anaphylactic or severe systemic response to immune Globulin (Human). Individuals with selective lgA deficiencies should not receive Gamma IV™, since these individuals may experience server reactions to the lgA which may be present.

Safety Warnings: The product should not be used if it is turbid. Solutions which have been frozen should not be used. Once opened, even if only partially used, vials should be discarded. IVIG should be administered only intravenously as the intramuscular and subcutaneous routes have not been evaluated.

Dosage and Administration: In general it is recommended that IVIG be administered by itself on an initial rate of 0.01 to 0.02 ml/kg body weighty/minute for 30 minutes, if well tolerated the rate may be gradually increased to a maximum of 0.08 ml/kg body weight/minute. IVIG is recommended to be given by a separate line by itself without mixing with other intravenous fluids or medications the patients might be receiving. IVIG is not compatible with saline. The dilution if required, IVIG may be diluted with 5% Dextrose in water.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1 and 14 years who had clinically diagnosed encephalitis on the basis of history of fever that lasted less than 14 days, altered consciousness with or without a history of new onset seizures with CSF finding of white cell count less than 1000 cells/mm3 with no organisms on Gram stain and a CSF: plasma glucose ratio > 40% admitted in Kanti Children's Hospital and BP Koirala Institute of Health Sciences, Nepal.

Exclusion Criteria:

* Asexual Plasmodium falciparum parasites in blood

  * Coma appears secondary to other systemic condition, eg hepatic failure, cardiac failure, toxins.
  * Patients who have documented antibiotic treatment before admission and in whom partially treated bacterial meningitis appears more likely than encephalitis
  * Children with simple febrile convulsions, defined as a single seizure lasting less than 15 minutes followed by full recovery of consciousness within 60 minutes.
  * Pregnant or breastfeeding females
  * Children with a GCS of 3/15, who were receiving artificial ventilation without signs of spontaneous respiration, and with absent oculocephalic reflex.

Ages: 1 Year to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Evidence of side effects of study drug such as infusion site reaction, diarrhea, rise in blood pressure and change in urinary output | Every 12 hours after administration of study drug upto discharge, which is on average eigth day (192 hours) of hospital admission
  Patients will be monitored for side effects such as infusion site reaction, diarrhea, rise in blood pressure (in mm Hg) and change in urinary output (in ml/Kg/hour) every 12 hours from first day of commencing treatment until until death or discharge. Patient on average are administered the study drug on the first day of admission. The study drug is administered daily for 5 days. Patients are discharged on an average on eighth day (192 hours) of hospital admission.

SECONDARY OUTCOMES:
Death or neurological sequelae | At the time of discharge, an expected average of eighth day of admission and again at 6 months after discharge
  At the time of discharge(expected average of eighth day of admission) or death: Time to death, to recover from coma, to sit independently, to stand independently, to walk at least 5m independently, and to leave hospital.
  At 6 months after discharge: history of further seizures, behavioral changes, evidence of recovery of neurological sequelae such as assessment of ability to sit independently, to stand independently, to walk at least 5 meters independently.

OTHER OUTCOMES:
Serum JEV PRNT50 level (immunological marker) | Measured at 3 time points: pre-treatment (just before first dose of study drug on first day), mid-treatment (just prior to fourth dose on fourth day) and post-treatment (one hour after fifth dose on fifth day).
  Pre-treatment was immediately prior to the first dose of study drug on the first day, mid-treatment was immediately prior to the 4th dose and post-treatment was 1hour after administering the fifth dose of the study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Solomon, MRCP, PhD, Study Chair — Director,Institute of Infection and Global Health, University of Liverpool, Apex Building, 8 West Derby Street, Liverpool, L69 7BE, UK , Head- Liverpool Brain Infection Group; Ajit Rayamajhi, MBBS, MD, Principal Investigator — Institute of Infection and Global Health, University of Liverpool, Liverpool, UK & Kanti Children's Hospital, Maharajgunj, Kathmandu, Nepal; Sam Nightingale, MRCP, Study Director — Institute of Infection and Global Health, University of Liverpool, Apex Building, 8 West Derby Street, Liverpool, L69 7BE, UK
Locations (2):
- Nepal (2):
  - Kanti Children's Hospital, Kathmandu, Bagmati
  - BP Koirala Institute of Health Sciences, Dharān, Koshi

REFERENCES:
- [Background] Solomon T, Dung NM, Kneen R, Gainsborough M, Vaughn DW, Khanh VT. Japanese encephalitis. J Neurol Neurosurg Psychiatry. 2000 Apr;68(4):405-15. doi: 10.1136/jnnp.68.4.405. No abstract available. PMID 10727474
- [Background] Tsai TF. New initiatives for the control of Japanese encephalitis by vaccination: minutes of a WHO/CVI meeting, Bangkok, Thailand, 13-15 October 1998. Vaccine. 2000 May 26;18 Suppl 2:1-25. doi: 10.1016/s0264-410x(00)00037-2. PMID 10821969
- [Background] Innis BL. Japanese encephalitis. In: Porterfield JS, editor. Exotic Viral Infections. London: Chapman & Hall; 1995. p. 147-74.
- [Background] Sumiyoshi H, Mori C, Fuke I, Morita K, Kuhara S, Kondou J, Kikuchi Y, Nagamatu H, Igarashi A. Complete nucleotide sequence of the Japanese encephalitis virus genome RNA. Virology. 1987 Dec;161(2):497-510. doi: 10.1016/0042-6822(87)90144-9. PMID 3686827
- [Background] Chambers TJ, Hahn CS, Galler R, Rice CM. Flavivirus genome organization, expression, and replication. Annu Rev Microbiol. 1990;44:649-88. doi: 10.1146/annurev.mi.44.100190.003245. No abstract available. PMID 2174669
- [Background] Gajanana A, Thenmozhi V, Samuel PP, Reuben R. A community-based study of subclinical flavivirus infections in children in an area of Tamil Nadu, India, where Japanese encephalitis is endemic. Bull World Health Organ. 1995;73(2):237-44. PMID 7743596
- [Background] HALSTEAD SB, GROSZ CR. Subclinical Japanese encephalitis. I. Infection of Americans with limited residence in Korea. Am J Hyg. 1962 Mar;75:190-201. No abstract available. PMID 13904014
- [Background] Solomon T, Dung NM, Kneen R, Thao le TT, Gainsborough M, Nisalak A, Day NP, Kirkham FJ, Vaughn DW, Smith S, White NJ. Seizures and raised intracranial pressure in Vietnamese patients with Japanese encephalitis. Brain. 2002 May;125(Pt 5):1084-93. doi: 10.1093/brain/awf116. PMID 11960897
- [Background] Solomon T, Kneen R, Dung NM, Khanh VC, Thuy TT, Ha DQ, Day NP, Nisalak A, Vaughn DW, White NJ. Poliomyelitis-like illness due to Japanese encephalitis virus. Lancet. 1998 Apr 11;351(9109):1094-7. doi: 10.1016/S0140-6736(97)07509-0. PMID 9660579
- [Background] Chen WR, Tesh RB, Rico-Hesse R. Genetic variation of Japanese encephalitis virus in nature. J Gen Virol. 1990 Dec;71 ( Pt 12):2915-22. doi: 10.1099/0022-1317-71-12-2915. PMID 2273391
- [Background] Chen WR, Rico-Hesse R, Tesh RB. A new genotype of Japanese encephalitis virus from Indonesia. Am J Trop Med Hyg. 1992 Jul;47(1):61-9. doi: 10.4269/ajtmh.1992.47.61. PMID 1322071
- [Background] Gould EA. Evolution of the Japanese serological group viruses. In: Mackenzie JS, Barrett AD, Deubel V, editors. Current Topics in Microbiology and Immunology: Japanese encephalitis and West Nile virus infections: Springer-Verlag; 2002. p. 391-404.
- [Background] Solomon T, Ni H, Beasley DW, Ekkelenkamp M, Cardosa MJ, Barrett AD. Origin and evolution of Japanese encephalitis virus in southeast Asia. J Virol. 2003 Mar;77(5):3091-8. doi: 10.1128/jvi.77.5.3091-3098.2003. PMID 12584335
- [Background] Shope RE. Concepts of control of Japanese encephalitis and dengue. Southeast Asian J Trop Med Public Health. 1997;28 Suppl 2:131-4. PMID 9561649
- [Background] Solomon T. Vaccines against Japanese encephalitis. In: Jong EC, Zuckerman JN, editors. Travelers' vaccines. Ontario, Canada: B.C. Decker; 2004. p. 219-56.
- [Background] Monath TP. Japanese encephalitis vaccines: current vaccines and future prospects. Curr Top Microbiol Immunol. 2002;267:105-38. doi: 10.1007/978-3-642-59403-8_6. PMID 12082985
- [Background] Bista MB, Banerjee MK, Shin SH, Tandan JB, Kim MH, Sohn YM, Ohrr HC, Tang JL, Halstead SB. Efficacy of single-dose SA 14-14-2 vaccine against Japanese encephalitis: a case control study. Lancet. 2001 Sep 8;358(9284):791-5. doi: 10.1016/s0140-6736(01)05967-0. PMID 11564484
- [Background] Solomon T, Dung NM, Wills B, Kneen R, Gainsborough M, Diet TV, Thuy TT, Loan HT, Khanh VC, Vaughn DW, White NJ, Farrar JJ. Interferon alfa-2a in Japanese encephalitis: a randomised double-blind placebo-controlled trial. Lancet. 2003 Mar 8;361(9360):821-6. doi: 10.1016/s0140-6736(03)12709-2. PMID 12642049
- [Background] Griffin DE. Immune responses to RNA-virus infections of the CNS. Nat Rev Immunol. 2003 Jun;3(6):493-502. doi: 10.1038/nri1105. PMID 12776209
- [Background] Irani DN. Central nervous system inflammation: can't live with it, can't live without it. Curr Opin Neurol. 2001 Jun;14(3):347-8. doi: 10.1097/00019052-200106000-00013. No abstract available. PMID 11371758
- [Background] Kimura T, Griffin DE. Extensive immune-mediated hippocampal damage in mice surviving infection with neuroadapted Sindbis virus. Virology. 2003 Jun 20;311(1):28-39. doi: 10.1016/s0042-6822(03)00110-7. PMID 12832200
- [Background] Hoke CH Jr, Vaughn DW, Nisalak A, Intralawan P, Poolsuppasit S, Jongsawas V, Titsyakorn U, Johnson RT. Effect of high-dose dexamethasone on the outcome of acute encephalitis due to Japanese encephalitis virus. J Infect Dis. 1992 Apr;165(4):631-7. doi: 10.1093/infdis/165.4.631. PMID 1313068
- [Background] Caramello P, Canta F, Balbiano R, Lipani F, Ariaudo S, De Agostini M, Calleri G, Boglione L, Di Caro A. Role of intravenous immunoglobulin administration in Japanese encephalitis. Clin Infect Dis. 2006 Dec 15;43(12):1620-1. doi: 10.1086/509644. No abstract available. PMID 17109300
- [Background] Agrawal AG, Petersen LR. Human immunoglobulin as a treatment for West Nile virus infection. J Infect Dis. 2003 Jul 1;188(1):1-4. doi: 10.1086/376871. Epub 2003 Jun 23. No abstract available. PMID 12825164
- [Background] Burke DS, Lorsomrudee W, Leake CJ, Hoke CH, Nisalak A, Chongswasdi V, Laorakpongse T. Fatal outcome in Japanese encephalitis. Am J Trop Med Hyg. 1985 Nov;34(6):1203-10. doi: 10.4269/ajtmh.1985.34.1203. PMID 3010752
- [Background] Solomon T, Thao LT, Dung NM, Kneen R, Hung NT, Nisalak A, Vaughn DW, Farrar J, Hien TT, White NJ, Cardosa MJ. Rapid diagnosis of Japanese encephalitis by using an immunoglobulin M dot enzyme immunoassay. J Clin Microbiol. 1998 Jul;36(7):2030-4. doi: 10.1128/JCM.36.7.2030-2034.1998. PMID 9650956
- [Background] Solomon T, Vaughn DW. Pathogenesis and clinical features of Japanese encephalitis and West Nile virus infections. Curr Top Microbiol Immunol. 2002;267:171-94. doi: 10.1007/978-3-642-59403-8_9. No abstract available. PMID 12082989
- [Background] Burke DS, Nisalak A, Lorsomrudee W, Ussery MA, Laorpongse T. Virus-specific antibody-producing cells in blood and cerebrospinal fluid in acute Japanese encephalitis. J Med Virol. 1985 Nov;17(3):283-92. doi: 10.1002/jmv.1890170310. PMID 2999326
- [Background] Desai A, Shankar SK, Ravi V, Chandramuki A, Gourie-Devi M. Japanese encephalitis virus antigen in the human brain and its topographic distribution. Acta Neuropathol. 1995;89(4):368-73. doi: 10.1007/BF00309631. PMID 7610769
- [Background] Shankar SK, Rao TV, Mruthyunjayanna BP, Gourie Devi M, Deshpande DH. Autopsy study of brains during an epidemic of Japanese encephalitis in Karnataka. Indian J Med Res. 1983 Sep;78:431-40. No abstract available. PMID 6325338
- [Background] Li ZS, Hong SF, Gong NL. Immunohistochemical study on Japanese B encephalitis. Chin Med J (Engl). 1988 Oct;101(10):768-71. No abstract available. PMID 2855049
- [Background] Johnson RT, Burke DS, Elwell M, Leake CJ, Nisalak A, Hoke CH, Lorsomrudee W. Japanese encephalitis: immunocytochemical studies of viral antigen and inflammatory cells in fatal cases. Ann Neurol. 1985 Nov;18(5):567-73. doi: 10.1002/ana.410180510. PMID 3000282
- [Background] MIYAKE M. THE PATHOLOGY OF JAPANESE ENCEPHALITIS. A REVIEW. Bull World Health Organ. 1964;30(2):153-60. PMID 14153404
- [Background] Solomon T. Flavivirus encephalitis. N Engl J Med. 2004 Jul 22;351(4):370-8. doi: 10.1056/NEJMra030476. No abstract available. PMID 15269317
- [Background] McMinn PC. The molecular basis of virulence of the encephalitogenic flaviviruses. J Gen Virol. 1997 Nov;78 ( Pt 11):2711-22. doi: 10.1099/0022-1317-78-11-2711. No abstract available. PMID 9367356
- [Background] Doherty PC, Zinkernagel RM. T-cell-mediated immunopathology in viral infections. Transplant Rev. 1974;19(0):89-120. doi: 10.1111/j.1600-065x.1974.tb00129.x. No abstract available. PMID 4601807
- [Background] Rowell JF, Griffin DE. Contribution of T cells to mortality in neurovirulent Sindbis virus encephalomyelitis. J Neuroimmunol. 2002 Jun;127(1-2):106-14. doi: 10.1016/s0165-5728(02)00108-x. PMID 12044981
- [Background] Atrasheuskaya A, Petzelbauer P, Fredeking TM, Ignatyev G. Anti-TNF antibody treatment reduces mortality in experimental dengue virus infection. FEMS Immunol Med Microbiol. 2003 Jan 21;35(1):33-42. doi: 10.1111/j.1574-695X.2003.tb00646.x. PMID 12589955
- [Background] Liu T, Chambers TJ. Yellow fever virus encephalitis: properties of the brain-associated T-cell response during virus clearance in normal and gamma interferon-deficient mice and requirement for CD4+ lymphocytes. J Virol. 2001 Mar;75(5):2107-18. doi: 10.1128/JVI.75.5.2107-2118.2001. PMID 11160715
- [Background] Wang Y, Lobigs M, Lee E, Mullbacher A. CD8+ T cells mediate recovery and immunopathology in West Nile virus encephalitis. J Virol. 2003 Dec;77(24):13323-34. doi: 10.1128/jvi.77.24.13323-13334.2003. PMID 14645588
- [Background] Wang T, Town T, Alexopoulou L, Anderson JF, Fikrig E, Flavell RA. Toll-like receptor 3 mediates West Nile virus entry into the brain causing lethal encephalitis. Nat Med. 2004 Dec;10(12):1366-73. doi: 10.1038/nm1140. Epub 2004 Nov 21. PMID 15558055
- [Background] Diamond MS, Klein RS. West Nile virus: crossing the blood-brain barrier. Nat Med. 2004 Dec;10(12):1294-5. doi: 10.1038/nm1204-1294. No abstract available. PMID 15580248
- [Background] Chambers TJ, Diamond MS. Pathogenesis of flavivirus encephalitis. Adv Virus Res. 2003;60:273-342. doi: 10.1016/s0065-3527(03)60008-4. PMID 14689697
- [Background] Myint KS, Gibbons RV, Perng GC, Solomon T. Unravelling the neuropathogenesis of Japanese encephalitis. Trans R Soc Trop Med Hyg. 2007 Oct;101(10):955-6. doi: 10.1016/j.trstmh.2007.04.004. Epub 2007 Jun 4. PMID 17544469
- [Background] Glass WG, McDermott DH, Lim JK, Lekhong S, Yu SF, Frank WA, Pape J, Cheshier RC, Murphy PM. CCR5 deficiency increases risk of symptomatic West Nile virus infection. J Exp Med. 2006 Jan 23;203(1):35-40. doi: 10.1084/jem.20051970. Epub 2006 Jan 17. PMID 16418398
- [Background] Glass WG, Lim JK, Cholera R, Pletnev AG, Gao JL, Murphy PM. Chemokine receptor CCR5 promotes leukocyte trafficking to the brain and survival in West Nile virus infection. J Exp Med. 2005 Oct 17;202(8):1087-98. doi: 10.1084/jem.20042530. PMID 16230476
- [Background] Bhowmick S, Duseja R, Das S, Appaiahgiri MB, Vrati S, Basu A. Induction of IP-10 (CXCL10) in astrocytes following Japanese encephalitis. Neurosci Lett. 2007 Feb 27;414(1):45-50. doi: 10.1016/j.neulet.2006.11.070. Epub 2007 Jan 8. PMID 17287085
- [Background] Ghoshal A, Das S, Ghosh S, Mishra MK, Sharma V, Koli P, Sen E, Basu A. Proinflammatory mediators released by activated microglia induces neuronal death in Japanese encephalitis. Glia. 2007 Apr 1;55(5):483-96. doi: 10.1002/glia.20474. PMID 17203475
- [Background] Li Y, Fu L, Gonzales DM, Lavi E. Coronavirus neurovirulence correlates with the ability of the virus to induce proinflammatory cytokine signals from astrocytes and microglia. J Virol. 2004 Apr;78(7):3398-406. doi: 10.1128/jvi.78.7.3398-3406.2004. PMID 15016862
- [Background] Allan SM, Rothwell NJ. Inflammation in central nervous system injury. Philos Trans R Soc Lond B Biol Sci. 2003 Oct 29;358(1438):1669-77. doi: 10.1098/rstb.2003.1358. PMID 14561325
- [Background] Van Wagoner NJ, Benveniste EN. Interleukin-6 expression and regulation in astrocytes. J Neuroimmunol. 1999 Dec;100(1-2):124-39. doi: 10.1016/s0165-5728(99)00187-3. PMID 10695723
- [Background] Frei K, Malipiero UV, Leist TP, Zinkernagel RM, Schwab ME, Fontana A. On the cellular source and function of interleukin 6 produced in the central nervous system in viral diseases. Eur J Immunol. 1989 Apr;19(4):689-94. doi: 10.1002/eji.1830190418. PMID 2543584
- [Background] Morris MM, Dyson H, Baker D, Harbige LS, Fazakerley JK, Amor S. Characterization of the cellular and cytokine response in the central nervous system following Semliki Forest virus infection. J Neuroimmunol. 1997 Apr;74(1-2):185-97. doi: 10.1016/s0165-5728(96)00786-2. PMID 9119972
- [Background] Brett FM, Mizisin AP, Powell HC, Campbell IL. Evolution of neuropathologic abnormalities associated with blood-brain barrier breakdown in transgenic mice expressing interleukin-6 in astrocytes. J Neuropathol Exp Neurol. 1995 Nov;54(6):766-75. doi: 10.1097/00005072-199511000-00003. PMID 7595649
- [Background] Paul R, Koedel U, Winkler F, Kieseier BC, Fontana A, Kopf M, Hartung HP, Pfister HW. Lack of IL-6 augments inflammatory response but decreases vascular permeability in bacterial meningitis. Brain. 2003 Aug;126(Pt 8):1873-82. doi: 10.1093/brain/awg171. Epub 2003 Jun 23. PMID 12821529
- [Background] Abraham CS, Deli MA, Joo F, Megyeri P, Torpier G. Intracarotid tumor necrosis factor-alpha administration increases the blood-brain barrier permeability in cerebral cortex of the newborn pig: quantitative aspects of double-labelling studies and confocal laser scanning analysis. Neurosci Lett. 1996 Apr 19;208(2):85-8. doi: 10.1016/0304-3940(96)12546-5. PMID 8859896
- [Background] Munoz-Fernandez MA, Fresno M. The role of tumour necrosis factor, interleukin 6, interferon-gamma and inducible nitric oxide synthase in the development and pathology of the nervous system. Prog Neurobiol. 1998 Oct;56(3):307-40. doi: 10.1016/s0301-0082(98)00045-8. PMID 9770242
- [Background] Griffin DE, Hardwick JM. Perspective: virus infections and the death of neurons. Trends Microbiol. 1999 Apr;7(4):155-60. doi: 10.1016/s0966-842x(99)01470-5. PMID 10217830
- [Background] Winter PM, Dung NM, Loan HT, Kneen R, Wills B, Thu le T, House D, White NJ, Farrar JJ, Hart CA, Solomon T. Proinflammatory cytokines and chemokines in humans with Japanese encephalitis. J Infect Dis. 2004 Nov 1;190(9):1618-26. doi: 10.1086/423328. Epub 2004 Sep 29. PMID 15478067
- [Background] Solomon T, Dung NM, Vaughn DW, Kneen R, Thao LT, Raengsakulrach B, Loan HT, Day NP, Farrar J, Myint KS, Warrell MJ, James WS, Nisalak A, White NJ. Neurological manifestations of dengue infection. Lancet. 2000 Mar 25;355(9209):1053-9. doi: 10.1016/S0140-6736(00)02036-5. PMID 10744091
- [Background] Leis AA, Stokic DS, Polk JL, Dostrow V, Winkelmann M. A poliomyelitis-like syndrome from West Nile virus infection. N Engl J Med. 2002 Oct 17;347(16):1279-80. doi: 10.1056/NEJM2002c021587. Epub 2002 Sep 23. No abstract available. PMID 12270971
- [Background] Solomon T, Winter PM. Neurovirulence and host factors in flavivirus encephalitis--evidence from clinical epidemiology. Arch Virol Suppl. 2004;(18):161-70. doi: 10.1007/978-3-7091-0572-6_14. PMID 15119771
- [Background] German AC, Myint KS, Mai NT, Pomeroy I, Phu NH, Tzartos J, Winter P, Collett J, Farrar J, Barrett A, Kipar A, Esiri MM, Solomon T. A preliminary neuropathological study of Japanese encephalitis in humans and a mouse model. Trans R Soc Trop Med Hyg. 2006 Dec;100(12):1135-45. doi: 10.1016/j.trstmh.2006.02.008. Epub 2006 Jun 30. PMID 16814333
- [Background] Ravi V, Parida S, Desai A, Chandramuki A, Gourie-Devi M, Grau GE. Correlation of tumor necrosis factor levels in the serum and cerebrospinal fluid with clinical outcome in Japanese encephalitis patients. J Med Virol. 1997 Feb;51(2):132-6. PMID 9021544
- [Background] Singh A, Kulshreshtha R, Mathur A. Secretion of the chemokine interleukin-8 during Japanese encephalitis virus infection. J Med Microbiol. 2000 Jul;49(7):607-612. doi: 10.1099/0022-1317-49-7-607. PMID 10882085
- [Background] Iwamoto M, Jernigan DB, Guasch A, Trepka MJ, Blackmore CG, Hellinger WC, Pham SM, Zaki S, Lanciotti RS, Lance-Parker SE, DiazGranados CA, Winquist AG, Perlino CA, Wiersma S, Hillyer KL, Goodman JL, Marfin AA, Chamberland ME, Petersen LR; West Nile Virus in Transplant Recipients Investigation Team. Transmission of West Nile virus from an organ donor to four transplant recipients. N Engl J Med. 2003 May 29;348(22):2196-203. doi: 10.1056/NEJMoa022987. PMID 12773646
- [Background] Chabas D, Baranzini SE, Mitchell D, Bernard CC, Rittling SR, Denhardt DT, Sobel RA, Lock C, Karpuj M, Pedotti R, Heller R, Oksenberg JR, Steinman L. The influence of the proinflammatory cytokine, osteopontin, on autoimmune demyelinating disease. Science. 2001 Nov 23;294(5547):1731-5. doi: 10.1126/science.1062960. PMID 11721059
- [Background] Lock C, Hermans G, Pedotti R, Brendolan A, Schadt E, Garren H, Langer-Gould A, Strober S, Cannella B, Allard J, Klonowski P, Austin A, Lad N, Kaminski N, Galli SJ, Oksenberg JR, Raine CS, Heller R, Steinman L. Gene-microarray analysis of multiple sclerosis lesions yields new targets validated in autoimmune encephalomyelitis. Nat Med. 2002 May;8(5):500-8. doi: 10.1038/nm0502-500. PMID 11984595
- [Background] Solomon T. Japanese encephalitis: Clinical features & pathogenesis. 55th Annual Meeting of the American Society of Tropical Medicine and Hygiene; 2006; Atlanta, Georgia; 2006.
- [Background] Edelman R, Schneider RJ, Vejjajiva A, Pornpibul R, Voodhikul P. Persistence of virus-specific IgM and clinical recovery after Japanese encephalitis. Am J Trop Med Hyg. 1976 Sep;25(5):733-8. doi: 10.4269/ajtmh.1976.25.733. PMID 183556
- [Background] Burke DS, Nisalak A, Ussery MA, Laorakpongse T, Chantavibul S. Kinetics of IgM and IgG responses to Japanese encephalitis virus in human serum and cerebrospinal fluid. J Infect Dis. 1985 Jun;151(6):1093-9. doi: 10.1093/infdis/151.6.1093. PMID 2987367
- [Background] Kumar R, Mathur A, Kumar A, Sharma S, Chakraborty S, Chaturvedi UC. Clinical features & prognostic indicators of Japanese encephalitis in children in Lucknow (India). Indian J Med Res. 1990 Sep;91:321-7. PMID 2176644
- [Background] Libraty DH, Nisalak A, Endy TP, Suntayakorn S, Vaughn DW, Innis BL. Clinical and immunological risk factors for severe disease in Japanese encephalitis. Trans R Soc Trop Med Hyg. 2002 Mar-Apr;96(2):173-8. doi: 10.1016/s0035-9203(02)90294-4. PMID 12055808
- [Background] Bista MB, Shrestha JM. Epidemiological situation of Japanese encephalitis in Nepal. JNMA J Nepal Med Assoc. 2005 Apr-Jun;44(158):51-6. PMID 16554872
- [Background] Rayamajhi A, Singh R, Prasad R, Khanal B, Singhi S. Clinico-laboratory profile and outcome of Japanese encephalitis in Nepali children. Ann Trop Paediatr. 2006 Dec;26(4):293-301. doi: 10.1179/146532806X152818. PMID 17132294
- [Background] Tandan JB, Ohrr H, Sohn YM, Yoksan S, Ji M, Nam CM, Halstead SB. Single dose of SA 14-14-2 vaccine provides long-term protection against Japanese encephalitis: a case-control study in Nepalese children 5 years after immunization. drjbtandan@yahoo.com. Vaccine. 2007 Jun 28;25(27):5041-5. doi: 10.1016/j.vaccine.2007.04.052. Epub 2007 May 8. PMID 17521781
- [Background] Pant GR. A serological survey of pigs, horses, and ducks in Nepal for evidence of infection with Japanese encephalitis virus. Ann N Y Acad Sci. 2006 Oct;1081:124-9. doi: 10.1196/annals.1373.013. PMID 17135501
- [Background] Leung DY, Burns JC, Newburger JW, Geha RS. Reversal of lymphocyte activation in vivo in the Kawasaki syndrome by intravenous gammaglobulin. J Clin Invest. 1987 Feb;79(2):468-72. doi: 10.1172/JCI112835. PMID 2433307
- [Background] Clarkson SB, Bussel JB, Kimberly RP, Valinsky JE, Nachman RL, Unkeless JC. Treatment of refractory immune thrombocytopenic purpura with an anti-Fc gamma-receptor antibody. N Engl J Med. 1986 May 8;314(19):1236-9. doi: 10.1056/NEJM198605083141907. No abstract available. PMID 2939345
- [Background] Buchwald B, Ahangari R, Weishaupt A, Toyka KV. Intravenous immunoglobulins neutralize blocking antibodies in Guillain-Barre syndrome. Ann Neurol. 2002 Jun;51(6):673-80. doi: 10.1002/ana.10205. PMID 12112071
- [Background] Quartier P, Foray S, Casanova JL, Hau-Rainsard I, Blanche S, Fischer A. Enteroviral meningoencephalitis in X-linked agammaglobulinemia: intensive immunoglobulin therapy and sequential viral detection in cerebrospinal fluid by polymerase chain reaction. Pediatr Infect Dis J. 2000 Nov;19(11):1106-8. doi: 10.1097/00006454-200011000-00020. No abstract available. PMID 11099099
- [Background] Spector SA, Gelber RD, McGrath N, Wara D, Barzilai A, Abrams E, Bryson YJ, Dankner WM, Livingston RA, Connor EM. A controlled trial of intravenous immune globulin for the prevention of serious bacterial infections in children receiving zidovudine for advanced human immunodeficiency virus infection. Pediatric AIDS Clinical Trials Group. N Engl J Med. 1994 Nov 3;331(18):1181-7. doi: 10.1056/NEJM199411033311802. PMID 7935655
- [Background] Rodriguez WJ, Gruber WC, Welliver RC, Groothuis JR, Simoes EA, Meissner HC, Hemming VG, Hall CB, Lepow ML, Rosas AJ, Robertsen C, Kramer AA. Respiratory syncytial virus (RSV) immune globulin intravenous therapy for RSV lower respiratory tract infection in infants and young children at high risk for severe RSV infections: Respiratory Syncytial Virus Immune Globulin Study Group. Pediatrics. 1997 Mar;99(3):454-61. doi: 10.1542/peds.99.3.454. PMID 9041304
- [Background] Keller MA, Stiehm ER. Passive immunity in prevention and treatment of infectious diseases. Clin Microbiol Rev. 2000 Oct;13(4):602-14. doi: 10.1128/CMR.13.4.602. PMID 11023960
- [Background] Levine B, Hardwick JM, Trapp BD, Crawford TO, Bollinger RC, Griffin DE. Antibody-mediated clearance of alphavirus infection from neurons. Science. 1991 Nov 8;254(5033):856-60. doi: 10.1126/science.1658936.
- [Background] Griffin DE, Ubol S, Despres P, Kimura T, Byrnes A. Role of antibodies in controlling alphavirus infection of neurons. Curr Top Microbiol Immunol. 2001;260:191-200. doi: 10.1007/978-3-662-05783-4_10. No abstract available. PMID 11443874
- [Background] Murali-Krishna K, Ravi V, Manjunath R. Protection of adult but not newborn mice against lethal intracerebral challenge with Japanese encephalitis virus by adoptively transferred virus-specific cytotoxic T lymphocytes: requirement for L3T4+ T cells. J Gen Virol. 1996 Apr;77 ( Pt 4):705-14. doi: 10.1099/0022-1317-77-4-705. PMID 8627259
- [Background] Pan CH, Chen HW, Huang HW, Tao MH. Protective mechanisms induced by a Japanese encephalitis virus DNA vaccine: requirement for antibody but not CD8(+) cytotoxic T-cell responses. J Virol. 2001 Dec;75(23):11457-63. doi: 10.1128/JVI.75.23.11457-11463.2001. PMID 11689627
- [Background] Beasley DW, Li L, Suderman MT, Guirakhoo F, Trent DW, Monath TP, Shope RE, Barrett AD. Protection against Japanese encephalitis virus strains representing four genotypes by passive transfer of sera raised against ChimeriVax-JE experimental vaccine. Vaccine. 2004 Sep 9;22(27-28):3722-6. doi: 10.1016/j.vaccine.2004.03.027. PMID 15315852
- [Background] Konishi E, Ajiro N, Nukuzuma C, Mason PW, Kurane I. Comparison of protective efficacies of plasmid DNAs encoding Japanese encephalitis virus proteins that induce neutralizing antibody or cytotoxic T lymphocytes in mice. Vaccine. 2003 Sep 8;21(25-26):3675-83. doi: 10.1016/s0264-410x(03)00382-7. PMID 12922097
- [Background] Kimura-Kuroda J, Yasui K. Protection of mice against Japanese encephalitis virus by passive administration with monoclonal antibodies. J Immunol. 1988 Nov 15;141(10):3606-10. PMID 2460542
- [Background] Zhang MJ, Wang MJ, Jiang SZ, Ma WY. Passive protection of mice, goats, and monkeys against Japanese encephalitis with monoclonal antibodies. J Med Virol. 1989 Oct;29(2):133-8. doi: 10.1002/jmv.1890290211. PMID 2557383
- [Background] Gupta AK, Lad VJ, Koshy AA. Protection of mice against experimental Japanese encephalitis virus infections by neutralizing anti-glycoprotein E monoclonal antibodies. Acta Virol. 2003;47(3):141-5. PMID 14658841
- [Background] Ben-Nathan D, Lustig S, Tam G, Robinzon S, Segal S, Rager-Zisman B. Prophylactic and therapeutic efficacy of human intravenous immunoglobulin in treating West Nile virus infection in mice. J Infect Dis. 2003 Jul 1;188(1):5-12. doi: 10.1086/376870. Epub 2003 Jun 23. PMID 12825165
- [Background] Diamond MS, Shrestha B, Marri A, Mahan D, Engle M. B cells and antibody play critical roles in the immediate defense of disseminated infection by West Nile encephalitis virus. J Virol. 2003 Feb;77(4):2578-86. doi: 10.1128/jvi.77.4.2578-2586.2003. PMID 12551996
- [Background] Kreil TR, Eibl MM. Pre- and postexposure protection by passive immunoglobulin but no enhancement of infection with a flavivirus in a mouse model. J Virol. 1997 Apr;71(4):2921-7. doi: 10.1128/JVI.71.4.2921-2927.1997. PMID 9060650
- [Background] Morrey JD, Siddharthan V, Olsen AL, Roper GY, Wang H, Baldwin TJ, Koenig S, Johnson S, Nordstrom JL, Diamond MS. Humanized monoclonal antibody against West Nile virus envelope protein administered after neuronal infection protects against lethal encephalitis in hamsters. J Infect Dis. 2006 Nov 1;194(9):1300-8. doi: 10.1086/508293. Epub 2006 Sep 22. PMID 17041857
- [Background] Morrey JD, Siddharthan V, Olsen AL, Wang H, Julander JG, Hall JO, Li H, Nordstrom JL, Koenig S, Johnson S, Diamond MS. Defining limits of treatment with humanized neutralizing monoclonal antibody for West Nile virus neurological infection in a hamster model. Antimicrob Agents Chemother. 2007 Jul;51(7):2396-402. doi: 10.1128/AAC.00147-07. Epub 2007 Apr 23. PMID 17452485
- [Background] Webb DB, Kendra JR, Gross E, Stamatakis JD. Infusion of intravenous immunoglobulin via implantable subcutaneous catheter. Lancet. 1991 Jun 29;337(8757):1617-8. doi: 10.1016/0140-6736(91)93323-2. No abstract available. PMID 1675753
- [Background] Imbach P. Immune thrombocytopenic purpura and intravenous immunoglobulin. Cancer. 1991 Sep 15;68(6 Suppl):1422-5. doi: 10.1002/1097-0142(19910915)68:6+3.0.co;2-5. PMID 1878840
- [Background] Dwyer JM. Manipulating the immune system with immune globulin. N Engl J Med. 1992 Jan 9;326(2):107-16. doi: 10.1056/NEJM199201093260206. No abstract available. PMID 1727218
- [Background] Sullivan KM, Kopecky KJ, Jocom J, Fisher L, Buckner CD, Meyers JD, Counts GW, Bowden RA, Peterson FB, Witherspoon RP, et al. Immunomodulatory and antimicrobial efficacy of intravenous immunoglobulin in bone marrow transplantation. N Engl J Med. 1990 Sep 13;323(11):705-12. doi: 10.1056/NEJM199009133231103. PMID 2167452
- [Background] Newburger JW, Takahashi M, Beiser AS, Burns JC, Bastian J, Chung KJ, Colan SD, Duffy CE, Fulton DR, Glode MP, et al. A single intravenous infusion of gamma globulin as compared with four infusions in the treatment of acute Kawasaki syndrome. N Engl J Med. 1991 Jun 6;324(23):1633-9. doi: 10.1056/NEJM199106063242305. PMID 1709446
- [Background] Ooi MH, Wong SC, Clear D, Perera D, Krishnan S, Preston T, Tio PH, Willison HJ, Tedman B, Kneen R, Cardosa MJ, Solomon T. Adenovirus type 21-associated acute flaccid paralysis during an outbreak of hand-foot-and-mouth disease in Sarawak, Malaysia. Clin Infect Dis. 2003 Mar 1;36(5):550-9. doi: 10.1086/367648. Epub 2003 Feb 14. PMID 12594634
- [Background] Chatterjee S, Chattopadhyay D, Bhattacharya MK, Mukherjee B. Serosurveillance for Japanese encephalitis in children in several districts of West Bengal, India. Acta Paediatr. 2004 Mar;93(3):390-3. PMID 15124845
- [Background] Planitzer CB, Modrof J, Kreil TR. West Nile virus neutralization by US plasma-derived immunoglobulin products. J Infect Dis. 2007 Aug 1;196(3):435-40. doi: 10.1086/519392. Epub 2007 Jun 18. PMID 17597458
- [Derived] Rayamajhi A, Nightingale S, Bhatta NK, Singh R, Kneen R, Ledger E, Bista KP, Lewthwaite P, Mahaseth C, Turtle L, Robinson JS, Galbraith SE, Wnek M, Johnson BW, Faragher B, Griffiths MJ, Solomon T. A preliminary randomized double blind placebo-controlled trial of intravenous immunoglobulin for Japanese encephalitis in Nepal. PLoS One. 2015 Apr 17;10(4):e0122608. doi: 10.1371/journal.pone.0122608. eCollection 2015. PMID 25886645